CLINICAL TRIAL: NCT02128854
Title: Tablet-Aided BehavioraL Intervention EffecT on Self-management Skills
Acronym: TABLETS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00021502; R03DK098489-01 (NIH)
Record Dates: First submitted 2014-04-18; First posted 2014-05-01 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2016-09

CONDITIONS: Diabetes Mellitus, Type 2; Diabetes Mellitus, Adult-Onset; Diabetes Mellitus, Non-Insulin-Dependent; Diabetes Mellitus, Noninsulin Dependent; Diabetes Mellitus, Type II
Keywords: Diabetes Mellitus, Type 2; Diabetes Mellitus, Adult-Onset; Diabetes Mellitus, Non-Insulin-Dependent; Diabetes Mellitus, Noninsulin Dependent; Diabetes Mellitus, Type II; African Americans; Blacks; Non-Hispanic Blacks; Randomized Control Trial; Controlled Clinical Trial; Behavioral Research; Behavioral Medicine
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Methods

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tablets Intervention (Experimental): Individuals randomized to this arm will receive: 1) peripheral devices for monitoring blood glucose, blood pressure, and weight; 2) 8 weekly tablet-delivered education and skills training sessions; 3) two booster sessions delivered via tablet-based videoconferencing at 3 and 6 months.
  Interventions: Behavioral: Tablets Intervention
- Usual Care (No Intervention): Apart from study visits, individuals randomized to the Usual Care group will receive usual care for diabetes management as provided by their primary care physician. The provider will be responsible for determining changes in the treatment regimen and determining the timing of follow-up visits for diabetes care. Between scheduled office encounters, contact will be initiated by the individual.

INTERVENTIONS:
Behavioral: Tablets Intervention — The TABLET intervention adds a novel tablet-based delivery mechanism to provide real-time videoconferencing education about diabetes self-management behaviors to high-risk, low-income African American (AA) adults with diabetes. Cardiovascular disease (CVD) knowledge/ information modules consist of materials developed from a CVD patient education booklet adapted from Maine Heart Center of Maine Health and supplemented by clinical guidelines to specifically address behavioral risk factors. Motivation/behavioral skills training modules consist of patient activation (asking questions to providers), patient empowerment (CVD responsibility contracts, flow charts for lab results), and behavioral skills training (self-monitoring, goal-setting).
  Arms: Tablets Intervention

SUMMARY:
The purpose of this project is two-fold: (1) to determine the feasibility of recruiting rural African American (AA) adults in South Carolina (SC) for assessing the usefulness of tablet-based resources in good diabetes self-management behaviors, and (2) to test a tablet-aided intervention for improving diabetes self-management behaviors

DETAILED DESCRIPTION:
The proposed study will assess the feasibility of recruitment of African American adults residing in rural South Carolina who will assist with improving the usability of tablet computers. In addition, we will implement a pilot trial of the TABLETS (Tablet-Aided BehavioraL intervention Effect on Self-management skills) intervention for diabetes, using motivational strategies, among rural African Americans. The proposed project is designed to address 3 important issues: recruitment for a hard-to-reach population, utility of technology-enabled intervention, and development of a tablet-aided intervention tailored to understand best practices for diabetes self-management

ELIGIBILITY:
Inclusion Criteria:

* Age ≥45 years
* Clinical diagnosis of diabetes with HbA1c ≥8% and either diagnosis of hyperlipidemia with LDL >100mg/dL or hypertension with BP >140/80mmHg
* Self-identified as African American
* Residence in a 4G cellular service area
* Able to communicate in English

Exclusion Criteria:

* Cognitive impairment
* Active alcohol or drug abuse/dependency
* Acute decompensation of chronic conditions precluding participation
* Participation in other diabetes clinical trials
* A life expectancy <6 months

Ages: 45 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-08-14 (Actual); Primary Completion 2016-07-26 (Actual); Study Completion 2016-08-31 (Actual)

PRIMARY OUTCOMES:
Self-Monitoring Behavior Using the Summary of Diabetes Self-Care Activities | 6 months post-randomization
  This will be done to assess self-management behaviors for diabetes.
Physical Activity Score on the Global Physical Activity Questionnaire | 6 months post-randomization
  Information will be collected to assess physical activity in three domains and sedentary behaviors.
Medication Adherence on the Morisky Medication Adherence Scale | 6 months post-randomization
  Scale will be used to assess specific medication-taking behaviors.
Diet Score on the Rapid Eating and Activity Assessment for Participants | 6 months post-randomization
  Dietary intake will be assessed.

SECONDARY OUTCOMES:
Glycosylated Hemoglobin A1c (HbA1c) | 6 months post-randomization
  Blood specimens (10cc of blood) will be obtained at baseline, 2, and 6-month visits for HbA1c.
Low-Density Lipoprotein Cholesterol (LDL-c) | 6 months post-randomization
  Blood specimens (10cc of blood) will be obtained at baseline, 2, and 6-month visits for non-fasting lipids.
Blood Pressure | 6 months post-randomization
  Blood pressure (BP) readings will be obtained using automated BP monitors. The device will be programmed to take 3 readings at 2 minute intervals, and give an average of the 3 BP readings.
Cardiovascular Disease (CVD) Risk Using the Framingham Risk Score | 6 months post-randomization
  This score will be used to estimate the 10-year risk for coronary heart disease outcomes (i.e., heart attack, death) according to 7 factors (age, gender, total cholesterol, high-density lipoprotein cholesterol, systolic blood pressure, high blood pressure medication use, and smoking status).
Quality of Life Using the Medical Outcomes Study Short Form | 6 months post-randomization
  We will obtain summary physical and mental health quality of life scores.

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl P Lynch, MD, MPH, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans to share IPD during the analysis phase.

REFERENCES:
- [Background] Lynch CP, Williams JS, J Ruggiero K, G Knapp R, Egede LE. Tablet-Aided BehavioraL intervention EffecT on Self-management skills (TABLETS) for Diabetes. Trials. 2016 Mar 22;17:157. doi: 10.1186/s13063-016-1243-2. PMID 27005766
- See also: Protocol paper — https://trialsjournal.biomedcentral.com/articles/10.1186/s13063-016-1243-2